CLINICAL TRIAL: NCT04619550
Title: Gait and Residual Pain at Different Physical Activity Intensities in High Tibial Osteotomy Patients and Healthy Controls
Brief Title: Gait, Pain and Physical Activity After HTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Winchester (Other)
Collaborators: RTI Surgical Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BLS/19/07
Record Dates: First submitted 2020-10-16; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis, Knee; Orthopedic Disorder
MeSH Terms: conditions — Osteoarthritis, Knee; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise intensity (Other): Jogging or walking at RPE 9, 11, 13, and 15
  Interventions: Other: High tibial osteotomy

INTERVENTIONS:
Other: High tibial osteotomy — Realignment surgery

SUMMARY:
This study aims to investigate the relationship between pain, gait and activity intensity in HTO patients that are healed and have had their fixation plate removed.

Inclusion criteria are: unilateral HTO with no concurrent procedure performed, fixation plate has since been removed, no subsequent operations performed on the lower limbs (hips to feet). Control participants will be recruited through local advertisements in and around the University of Winchester. Inclusion criteria for the control subjects are: no current pain in the lower limbs, no previous surgery on the lower limbs. Control subjects will also be age-matched to the HTO group.

Knee function and pain scores will first be assessed through the implementation of a Knee Osteoarthritis Outcome Score, a Visual Analogue Scale, and a further pain intensity scale. Once this has been done, resting heart rate (HR) and body mass index (BMI) will also be measured as part of the completion of a Physical Activity Readiness Questionnaire (PAR-Q). A G-Walk gait analysis sensor, which has been validated for use in clinical settings, will then be attached to participants in order to measure spatiotemporal gait parameters during testing.

Each participant will then conduct a series of four walking and four jogging test protocols, each lasting three minutes, on a flat treadmill. The intensity at which the participant must walk or jog during each test will be self-regulated and determined by a rating of perceived exertion (RPE) of 9, 11, 13 or 15 on a 6-20 Borg scale. All participants will be verbally anchored to the Borg scale before conducting the first walk/jog test. The order in which the tests are performed will be randomised in advance of each test session. Half way through each test (90 seconds), participants will be presented with a VAS and pain intensity scale to indicate the current level of pain they are experiencing in their knee. At this stage, they will also be asked to confirm that they are still maintaining the target RPE of that particular test. Once a test is finished, participants will complete another VAS and pain intensity scale and rest in a seated position until their heart rate returns to their pre-determined resting level before the next test commences. The leg for which healthy controls report pain levels will be chosen randomly prior to the test session.

DETAILED DESCRIPTION:
This study aims to investigate the relationship between pain, gait and activity intensity in HTO patients that are healed and have had their fixation plate removed.

Inclusion criteria are: unilateral HTO with no concurrent procedure performed, fixation plate has since been removed, no subsequent operations performed on the lower limbs (hips to feet). Control participants will be recruited through local advertisements in and around the University of Winchester. Inclusion criteria for the control subjects are: no current pain in the lower limbs, no previous surgery on the lower limbs. Control subjects will also be age-matched to the HTO group.

Knee function and pain scores will first be assessed through the implementation of a Knee Osteoarthritis Outcome Score, a Visual Analogue Scale, and a further pain intensity scale. Once this has been done, resting heart rate (HR) and body mass index (BMI) will also be measured as part of the completion of a Physical Activity Readiness Questionnaire (PAR-Q). A G-Walk gait analysis sensor, which has been validated for use in clinical settings, will then be attached to participants in order to measure spatiotemporal gait parameters during testing.

Each participant will then conduct a series of four walking and four jogging test protocols, each lasting three minutes, on a flat treadmill. The intensity at which the participant must walk or jog during each test will be self-regulated and determined by a rating of perceived exertion (RPE) of 9, 11, 13 or 15 on a 6-20 Borg scale. All participants will be verbally anchored to the Borg scale before conducting the first walk/jog test. The order in which the tests are performed will be randomised in advance of each test session. Half way through each test (90 seconds), participants will be presented with a VAS and pain intensity scale to indicate the current level of pain they are experiencing in their knee. At this stage, they will also be asked to confirm that they are still maintaining the target RPE of that particular test. Once a test is finished, participants will complete another VAS and pain intensity scale and rest in a seated position until their heart rate returns to their pre-determined resting level before the next test commences. The leg for which healthy controls report pain levels will be chosen randomly prior to the test session.

ELIGIBILITY:
Inclusion Criteria:

* Experimental group:

Previously undergone unilateral medial opening wedge high tibial osteotomy with no simultaneous procedures (other than arthroscopy), performed by one of 3 different surgeons

Plate since removed

No conversion to arthroplasty since the osteotomy

* Control group:

Age-matched to experimental group

Never previously undergone any form of lower limb surgery

Exclusion Criteria:

* Experimental group:

Undergone other procedures simultaneous to the osteotomy

Plate in-situ

* Control group:

Previously undergone lower limb surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Spatiotemporal parameters of gait | 9 months recruitment - 2 hours data collection per participant
  Steps, cadence, speed (etc) measured using G-Walk wireless inertial sensor
Self-reported pain questionnaire | 9 months recruitment - 2 hours data collection per participant
  Visual analogues scale (0-10, where 0 = no pain and 10 = the worst imaginable pain)

SECONDARY OUTCOMES:
Self-reported knee function questionnaire | 9 months recruitment - 2 hours data collection per participant
  Knee Osteoarthritis Outcome Score validated questionnaire (score /100, where higher number = better knee function)

CONTACTS AND LOCATIONS:
Overall Officials: James Belsey, MA, Principal Investigator — University of Winchester
Locations (1):
- University of Winchester, Winchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No